CLINICAL TRIAL: NCT00366873
Title: Evaluation of Mineral Absorption in Infants Fed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Carol Berseth, MD, Mead Johnson
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 3374-1151
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Infant; Term

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): cow-milk based infant formula
  Interventions: Procedure: Calcium absorption
- 2 (Experimental): cow-milk based infant formula with prebiotics
  Interventions: Procedure: Calcium absorption

INTERVENTIONS:
Procedure: Calcium absorption — formula with or without prebiotics

SUMMARY:
The purpose of this study is to measure calcium absorption in infants fed formula with and without prebiotics.

DETAILED DESCRIPTION:
Infants will be fed formula and blood drawn and urine collected to measure calcium absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infants

Exclusion Criteria:

* Breast fed infants
* Use of vitamin/mineral supplements
* Currently on medication

Ages: 56 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Calcium absorption | 14 days

SECONDARY OUTCOMES:
Vitamin D levels | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: James Heubi, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Fomon Infant Nutrition Unit, Coralville, Iowa
  - Pediatric Clinical Trials Unit, Louisville, Kentucky
  - The Center for Human Nutrition, Omaha, Nebraska
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Research and Nutrition Center, Houston, Texas